CLINICAL TRIAL: NCT02326805
Title: Phase II Randomized, Placebo-Controlled Trial of PROSTVAC (PSA-TRICOM) in Patients With Clinically Localized Prostate Cancer Undergoing Active Surveillance
Brief Title: PROSTVAC (PSA-TRICOM) in Preventing Disease Progression in Patients With Localized Prostate Cancer Undergoing Active Surveillance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCI-2014-02556; NCI-2014-02556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AZ027; HHSN2612012000311; N01-CN-2012-00031; 1410547210 (Other: Banner University Medical Center - Tucson); UAZ2014-03-01 (Other: DCP); N01CN00031 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Stage I Prostate Adenocarcinoma AJCC v7; Stage II Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — PROSTVAC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (rilimogene-galvacirepvec) (Experimental): Patients receive rilimogene-galvacirepvec SC at baseline and on days 14, 28, 56, 84, 112, and 140.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Rilimogene Galvacirepvec
- Arm II (placebo) (Placebo Comparator): Patients receive placebo SC at baseline and on days 14, 28, 56, 84, 112, and 140.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given SC
  Arms: Arm II (placebo)
Biological: Rilimogene Galvacirepvec — Given SC
  Other Names: PROSTVAC; Prostvac-V; Recombinant Vaccinia-PSA(L155)-TRICOM Vaccine; Recombinant Vaccinia-PSA(L155)/TRICOM; Recombinant Vaccinia-PSA(L155)/TRICOM Vaccine; rVaccinia-Prostate-Specific Antigen/TRICOM Vaccine; rVaccinia-PSA(L155)-TRICOM Vaccine
  Arms: Arm I (rilimogene-galvacirepvec)

SUMMARY:
This randomized phase II trial studies how well PROSTVAC (prostate-specific antigen [PSA]-TRICOM) works in preventing disease progression in patients with prostate cancer undergoing active surveillance. Vaccines made from a person's tumor cells may help the body build an effective immune response to kill tumor cells that express PSA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of rilimogene-galvacirepvec (PROSTVAC) on the change (from pre to post-intervention) in CD8+ positive cells in the stroma adjacent to tumor and within the malignant portion of the prostate biopsies.

II. To determine the effect of PROSTVAC on the change in CD4+ positive cells in the stroma adjacent to tumor and within the malignant portion of the prostate biopsies.

SECONDARY OBJECTIVES:

I. To assess the effect of PROSTVAC on PD-L1 positive cells in the stroma adjacent to tumor and within the malignant portion of the prostate biopsies.

II. To assess the correlation between the change in CD8+ and the change in PSA. III. To assess the effect of PROSTVAC on CD8+, CD4+, and PD-L1 positive cells in the benign portion of the prostate biopsies.

IV. To assess the effect of PROSTVAC on the change in PSA. V. To assess the effect of PROSTVAC on tumor grade (Gleason score). VI. To assess the effect of PROSTVAC on tumor extent (percent of positive random biopsy cores).

VII. To compare the proportion of men on the two study arms with no cancer on post-intervention biopsy.

VIII. To assess the effect of PROSTVAC on the size of the dominant lesion on magnetic resonance imaging (MRI) (largest histopathologically confirmed lesion) in the subgroup of patients with MRIs pre and postintervention.

IX. To assess the effect of PROSTVAC on circulating 15-Mer PSA-specific, MUC-1 and Brachyury-specific T cells.

X. To assess the effect of PROSTVAC on soluble antibodies to tumor-associated antigens.

XI. To assess the immunologic effects of PROSTVAC in prostate tissue using multiplex immunofluorescence.

XII. To assess the safety and feasibility of PROSTVAC in the active surveillance population.

XIII. To assess the effect of PROSTVAC on lower urinary tract symptoms (LUTS) in the active surveillance population.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive rilimogene-galvacirepvec subcutaneously (SC) at baseline and on days 14, 28, 56, 84, 112, and 140.

ARM II: Patients receive placebo SC at baseline and on days 14, 28, 56, 84, 112, and 140.

After completion of study treatment, patients are followed up for 30 days and then at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven (consisting of >= 10 tissue cores) adenocarcinoma of the prostate with cancer present in at least one biopsy core, either random or targeted, in the most recent biopsy

  * All prior biopsies must meet the following: =< 50% of the total number of random biopsy cores positive for cancer
  * Gleason score =< (3+4)
* Clinical stage =< T2a by digital rectal exam (DRE)
* Biopsies performed at outside institutions should have Gleason score confirmed at the study site by a genitourinary (GU) pathologist to ensure eligibility
* Pre-intervention biopsy tissue (most proximal to enrollment) with sufficient tumor tissue to cut 5-10 unstained slides confirmed to be available upon request
* Screening serum PSA < 20 ng/mL; for men treated with 5-alpha-reductase inhibitors (e.g., finasteride, dutasteride), PSA needs to be < 10 ng/mL
* Neutrophil count >= 1,200/mm^3 (>= 1.2 k/uL)
* Stable platelet count >= 75,000/mm^3 (>= 75 k/uL)
* Bilirubin =< 1.5 mg/dL (or =< 3.0 mg/dL for patients with Gilbert's syndrome)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 x ULN
* Karnofsky >= 70%
* Must agree to use medically acceptable barrier and/or chemical method of contraception while on study and for at least one month following the last vaccine injection; should a participant's partner become pregnant or suspect she is pregnant while the participant is participating in this study, the study physician should be informed immediately; in the event a participant's partner becomes pregnant, the study sponsor may request additional information regarding the course of the pregnancy and if the pregnancy is carried to term, the birth of the child (i.e., the outcome of the pregnancy)
* Ability to understand and the willingness to sign a written informed consent document
* No planned prostate biopsies during the intervention until after the post-intervention biopsy
* Men on stable doses of 5-alpha reductase inhibitors are eligible as long as there is no planned dose change while on study

Exclusion Criteria:

* Have had prior treatment for prostate cancer by surgery, irradiation, local ablative (i.e., cryosurgery or high-intensity focused ultrasound), or androgen-deprivation therapy
* Patients who have prostate cancer with distant metastases
* Have undergone treatment of hormone therapy, immunotherapy, chemotherapy and/or radiation for any malignancies within the past 2 years
* Uncontrolled intermittent illnesses or medical conditions which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient; such illnesses/conditions may include, but are not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Positive for human immunodeficiency virus (HIV) or active infections for hepatitis B, and/or hepatitis C, based on medical history
* Prior solid organ or bone marrow transplant
* Immunodeficiency or splenectomy
* Chronic immunosuppressive therapy within 30 days of screening
* Inflammatory eye disease requiring steroid treatment within 28 days of screening
* Chronic administration (defined as daily or every other day for continued use > 14 days) of systemic corticosteroids within 28 days of the first planned dose of PROSTVAC-V/F; use of inhaled steroids, nasal sprays, and topical creams for small body areas is allowed
* History of or active autoimmune disease including but not limited to autoimmune neutropenia, thrombocytopenia, or hemolytic anemia, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome; persons with vitiligo are not excluded; Persons with well-controlled autoimmune endocrinopathies, e.g., diabetes mellitus, Graves' disease, Hashimoto's thyroiditis, Addison's disease are not excluded; persons with well-controlled rheumatoid arthritis, psoriatic arthritis and polymyalgia rheumatica are not excluded
* Known allergy to eggs, egg products
* Prior or concurrent eczema or other eczemoid skin disorders or active skin condition (acute, chronic, or exfoliative) that disrupts the epidermis; persons with psoriasis are not excluded except in cases of:

  * any active lesion
  * any active lesion in the previous 6 months that required treatment, either systemic or topical
  * any prior episode, at any time, extensive enough or severe enough as to require systemic treatment
* Previous adverse reactions to smallpox vaccination
* Unable to avoid close contact or household contact with the following high-risk individuals for three weeks after the day 1 vaccination or until the vaccination site heals completely: (a) children =< 3 years of age, (b) pregnant or nursing women, (c) individuals with prior or concurrent extensive eczema or other eczemoid skin disorders, (d) individuals with other acute, chronic, or exfoliative skin condition, or (e) immunocompromised or immunosuppressed persons (by disease or therapy)
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition of PROSTVAC

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Parsons, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (7):
- United States (7):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Derived] Parsons JK, Pinto PA, Pavlovich CP, Uchio E, Kim HL, Nguyen MN, Gulley JL, Jamieson C, Hsu P, Wojtowicz M, Parnes H, Schlom J, Dahut WL, Madan RA, Donahue RN, Chow HS. A Randomized, Double-blind, Phase II Trial of PSA-TRICOM (PROSTVAC) in Patients with Localized Prostate Cancer: The Immunotherapy to Prevent Progression on Active Surveillance Study. Eur Urol Focus. 2018 Sep;4(5):636-638. doi: 10.1016/j.euf.2018.08.016. Epub 2018 Sep 7. PMID 30197041

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Started | 106 | 48
Completed | 103 | 47
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo) | Total
Number analyzed (Participants) | 106 | 48 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 64 (8) | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 106 | 48 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 98 | 45 | 143
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 5 | 12
  White | 91 | 43 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 106 | 48 | 154

OUTCOME MEASURES:

1. Primary Outcome: Change in CD8+ Positive Cells in the Stroma Adjacent to Tumor and Within the Malignant Portion of the Prostate Biopsies
Description: change (from pre to post-intervention) in CD8+ positive cells in the stroma adjacent to tumor and within the malignant portion of the prostate biopsies.
Time Frame: Baseline to up to 14 days after the last dose
Population: Participants with tumor present in tissue sections from both the pre and post-intervention biopsies
Measure: Mean (Standard Deviation); unit: number of positive cells per mm^2
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 72 | 28
number of positive cells per mm^2 | 12.2 (151.4) | -6.9 (154)

2. Primary Outcome: Change in CD4+ Positive Cells in the Stroma Adjacent to Tumor and Within the Malignant Portion of the Prostate Biopsies
Description: change (from pre to post-intervention) in CD4+ positive cells in the stroma adjacent to tumor and within the malignant portion of the prostate biopsies.
Time Frame: Baseline to up to 14 days after the last dose
Population: Participants with tumor present on the tissue sections from both the pre and post-intervention biopsies were included in the analysis
Measure: Mean (Standard Deviation); unit: number of positive cells per mm^2
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 69 | 28
number of positive cells per mm^2 | 4.6 (166.7) | 5.8 (261.1)

3. Secondary Outcome: Change in PD-L1 Positive Cells in the Stroma Adjacent to Tumor and Within the Malignant Portion of the Prostate Biopsies
Description: Change (from pre to post-intervention) in PD-L1 positive cells in the stroma adjacent to tumor and within the malignant portion of the prostate biopsies
Time Frame: Baseline to 6 months post-intervention
Population: Data were not obtained.
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Prostate-specific Antigen (PSA)
Description: Change (from baseline to 6 months post-intervention) in prostate-specific antigen (PSA)
Time Frame: Baseline to 6 months post-intervention
Population: The initial protocol did not include participant follow-up at 6 months post-intervention. Participants with available PSA data at baseline and at 6 months post-intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 76 | 35
ng/ml | 0.26 (2.36) | -0.66 (3.49)

5. Secondary Outcome: Change in CD8+ Positive Cells in the Benign Portion of the Prostate Biopsies
Description: Change (from pre to post-intervention) in CD8+ positive cells in the benign portion of the prostate biopsies
Time Frame: Baseline to up to 14 days after the last dose
Population: Participants with benign tissue present in tissue sections from both the pre and post-intervention biopsies were included in the analysis.
Measure: Mean (Standard Deviation); unit: number of positive cells per mm^2
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 74 | 34
number of positive cells per mm^2 | 7.22 (202.94) | 45.25 (198.25)

6. Secondary Outcome: Change in CD4+ Positive Cells in the Benign Portion of the Prostate Biopsies
Description: Change (from pre to post-intervention) in CD4+ positive cells in the benign portion of the prostate biopsies
Time Frame: Baseline to up to 14 days after the last dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of positive cells per mm^2
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 69 | 34
number of positive cells per mm^2 | 73.41 (287.74) | -19.75 (206.59)

7. Secondary Outcome: Change in PD-L1 Positive Cells in the Benign Portion of the Prostate Biopsies
Description: Change (from pre to post-intervention) in PD-L1 positive cells in the benign portion of the prostate biopsies
Time Frame: Baseline to up to 14 days after the last dose
Population: Data were not obtained.
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Tumor Grade Progression
Description: Assessed by the proportion of men with an increase in Gleason score to >= 4+3 from baseline to post-intervention biopsy. The Gleason score is determined by adding the two most common grades. The Gleason score usually ranges from 6 to 10. Higher numbers indicate a faster growing cancer that is more likely to spread.
Time Frame: Baseline to up to 14 days after the last dose
Population: The number of participants analyzed is different from the numbers provided in the Participant Flow Module because 2 participants in the placebo arm did not undergo the post-intervention biopsy to provide the data for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 106 | 46
Participants | 8 | 6

9. Secondary Outcome: Change in Tumor Extent
Description: Assessed by change (from pre to post-intervention) in percent positive random cores
Time Frame: Baseline to up to 14 days after the last dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of total cores
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 106 | 46
percentage of total cores | -1.7 (16.1) | 1.6 (15.2)

10. Secondary Outcome: Proportion of Men With no Cancer in the Post-intervention Biopsy
Description: Assessed by the proportion of patients with no cancer on the post-intervention biopsy
Time Frame: Up to 14 days after the last dose
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 106 | 46
Participants | 25 | 8

11. Secondary Outcome: Size of Dominant MRI Lesion
Description: The size of dominant MRI lesion.
Time Frame: Up to 14 days after the last dose
Population: Data were not collected.
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Circulating 15-Mer PSA-specific T Cells
Description: Change (from pre to post-intervention) in circulating 15-Mer PSA-specific T cells
Time Frame: Baseline to up to 14 days after the last dose
Population: Data were not collected.
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Soluble Antibodies to Tumor-associated Antigens
Description: Change (from pre to post-intervention) in soluble antibodies to tumor-associated antigens
Time Frame: Baseline to up to 14 days after the last dose
Population: Data were not collected.
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Immunologic Effects on the Target Organ Using Multiplex Immunofluorescence
Time Frame: Up to 14 days after the last dose
Population: Data were not collected.
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in International Prostate Symptom Score
Description: Change (from baseline to 6 months post-intervention) in International Prostate Symptom Score (IPSS). The IPSS score ranges from 0-35. Higher scores mean a worse symptom.
Time Frame: Baseline to up to 6 months post-intervention
Population: The initial protocol did not include participant follow-up at 6 months post-intervention. Participants with available IPSS data at baseline and at 6 months post-intervention were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
Number analyzed (Participants) | 58 | 30
score on a scale | -0.12 (4.67) | 0.87 (3.57)

ADVERSE EVENTS:
Time Frame: 30 days after the last study dose was given
Arm/Group | Arm I (Rilimogene-galvacirepvec) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/106 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/106 | 0/48
Other Adverse Events (participants affected / at risk) | 103/106 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Rilimogene-galvacirepvec) (N=106) | Arm II (Placebo) (N=48)
Fall (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Rilimogene-galvacirepvec) (N=106) | Arm II (Placebo) (N=48)
Diarrhea (Gastrointestinal disorders) | 10 | 6
Nausea (Gastrointestinal disorders) | 9 | 2
Fatigue (General disorders) | 43 | 14
Fever (General disorders) | 17 | 6
Flu like syndromes (Hepatobiliary disorders) | 63 | 30
Injection site reaction (General disorders) | 95 | 45
Upper respiratory infection (Infections and infestations) | 10 | 4
Bruising (Injury, poisoning and procedural complications) | 6 | 3
White blood cell decreased (Investigations) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 2
Renal and urinary disorders - others (Renal and urinary disorders) | 2 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 10 | 0
Headache (Nervous system disorders) | 23 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT02326805/Prot_SAP_ICF_001.pdf